CLINICAL TRIAL: NCT01258595
Title: Safety and Immunogenicity of High-Dose Trivalent Inactivated Influenza Vaccine in Adults 50 to 64 Years of Age
Brief Title: A Study of High-Dose Trivalent Inactivated Influenza Vaccine in Adults 50 to 64 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FIM09; UTN: U1111-1113-3648 (Other: WHO)
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Results first posted 2011-10-27 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
Keywords: Influenza; Trivalent Inactivated Influenza Vaccine; High-Dose Trivalent Inactivated Influenza Vaccine; Influenza vaccines
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-Dose Trivalent Inactivated Influenza Vaccine (Experimental)
  Interventions: Biological: High-Dose Trivalent Inactivated Influenza Vaccine
- Trivalent Inactivated Influenza Vaccine (Active Comparator)
  Interventions: Biological: Trivalent Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: High-Dose Trivalent Inactivated Influenza Vaccine — 0.5 mL Intramuscular
  Other Names: Fluzone® High-Dose
  Arms: High-Dose Trivalent Inactivated Influenza Vaccine
Biological: Trivalent Inactivated Influenza Vaccine — 0.5 mL, Intramuscular
  Other Names: Fluzone®
  Arms: Trivalent Inactivated Influenza Vaccine

SUMMARY:
The aim of the study is to generate data on key parameters associated with assessment of influenza vaccines in individuals 50-64 years of age

Primary Objective:

* To describe the immunogenicity of High-Dose Trivalent Inactivated Influenza Vaccine (TIV) compared to TIV.
* To describe the safety profile of High-Dose Trivalent Inactivated Influenza Vaccine, as assessed by solicited adverse reactions collected for 7 days post-vaccination, and unsolicited adverse events (including Serious Adverse Events and Adverse Events of Special Interests) collected between Visit 1 and Visit 2

DETAILED DESCRIPTION:
Participants will be randomized to receive one dose of either High-Dose Trivalent Inactivated Influenza Vaccine or Trivalent Inactivated Influenza Vaccine. They will be followed up for safety for one month post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 to 64 years (inclusive) on the day of vaccination
* Informed consent form has been signed and dated
* Medically stable
* Able to attend all scheduled visits and to comply with all trial procedures
* For a woman of childbearing potential, use of an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination

Exclusion Criteria:

* Known pregnancy, or a positive urine pregnancy test
* Currently breastfeeding a child
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Planned receipt of any vaccine in the 4 weeks following the trial vaccination (prior to the Visit 2 blood draw)
* Receipt of seasonal or pandemic influenza vaccine in the past 6 months
* Receipt of blood or blood-derived products in the past 3 months
* Systemic hypersensitivity to eggs, chicken proteins, or any of the vaccine components, or a history of a life-threatening reaction to the standard-dose Trivalent Inactivated Influenza Vaccine or a vaccine containing any of the same substances
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy
* Neoplastic disease or any hematologic malignancy
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination
* Personal history of Guillain-Barré Syndrome
* Self-reported seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Identified as employees of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members (i.e., immediate, husband, wife and their children, adopted or natural) of the employees or the Investigator

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (5):
- United States (5):
  - Idaho Falls, Idaho
  - Columbia, Maryland
  - Ellicott City, Maryland
  - Missoula, Montana
  - Cleveland, Ohio

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 15 November to 10 December 2010 in 4 clinical centers in the US.
Pre-assignment Details: A total of 300 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Fluzone® High-Dose Vaccine Group: Participants who received a single dose of Fluzone® High-Dose vaccine, containing 60 µg hemagglutinin on Day 0
- Fluzone® Vaccine Group: Participants who received a single dose of Fluzone® vaccine, containing 15 µg hemagglutinin on Day 0
Period: Overall Study
Arm/Group | Fluzone® High-Dose Vaccine Group | Fluzone® Vaccine Group
Started | 148 | 152
Completed | 147 | 151
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluzone® High-Dose Vaccine Group | Fluzone® Vaccine Group | Total
Number analyzed (Participants) | 148 | 152 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 148 | 152 | 300
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.6 (4.38) | 57.7 (4.14) | 57.7 (4.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 96 | 194
  Male | 50 | 56 | 106
Region of Enrollment [Number; unit: Participants]
  United States | 148 | 152 | 300

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Vaccine Antibodies Before and After Vaccination With Either Fluzone® High-Dose or Fluzone® Vaccine.
Description: Serum antibody titers to vaccine antigens were assessed by means of the hemagglutination inhibition (HAI) assay method.
Time Frame: Day 0 and Day 28 post-vaccination
Population: Serum antibody titers to vaccine antigens were assessed in the full analysis set population.
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution (1/dil)
Arm/Group | Fluzone® High-Dose Vaccine Group | Fluzone® Vaccine Group
Number analyzed (Participants) | 147 | 152
1/dilution (1/dil)
  A/H1N1: California - Pre-vaccination (N=147, 152) | 40.5 [30.0 to 54.5] | 28.8 [21.8 to 38.1]
  A/H3N2: Victoria - Pre-vaccination (N=147, 152) | 36.4 [28.0 to 47.4] | 41.4 [31.4 to 54.6]
  B: Brisbane - Pre-vaccination (N=147, 152) | 27.4 [22.4 to 33.6] | 28.9 [23.5 to 35.5]
  A/H1N1: California - Post-vaccination (N=145, 151) | 1067 [868 to 1312] | 745 [585 to 948]
  A/H3N2: Victoria - Post-vaccination (N = 145, 151) | 936 [745 to 1176] | 567 [459 to 699]
  B: Brisbane - Post-vaccination (N=145, 151) | 203 [171 to 241] | 127 [104 to 154]

2. Primary Outcome: Geometric Mean of Individual Titer Ratios (GMTRs) of Vaccine Antibodies Before and After Vaccination With Either Fluzone® High-Dose or Fluzone® Vaccine
Description: Serum antibody titers to vaccine antigens were assessed by means of the hemagglutination inhibition (HAI) assay method.
Time Frame: Day 0 and Day 28 Post-vaccination
Population: Serum antibody titers to vaccine antigens were assessed in the full analysis set population.
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution (1/dil)
Arm/Group | Fluzone® High-Dose Vaccine Group | Fluzone® Vaccine Group
Number analyzed (Participants) | 145 | 151
1/dilution (1/dil)
  A/H1N1: California | 21.8 [16.1 to 29.6] | 21.2 [15.8 to 28.4]
  A/H3N2: Victoria | 22.0 [17.2 to 28.1] | 12.0 [9.21 to 15.5]
  B: Brisbane | 6.27 [5.16 to 7.62] | 3.91 [3.17 to 4.83]

3. Primary Outcome: Percentage of Participants With Seroconversion After Vaccination With Either Fluzone® High-Dose or Fluzone® Vaccine
Description: Seroconversion: For participants with a Day 0 (pre-vaccination) titer < 10 (1/dilution [1/dil]) a titer ≥ 40 (1/dil), and for participants with a Day 0 titer ≥ 10 (1/dil) a ≥ 4 fold increase of titer on Day 28.
  Serum antibody titers were assessed by means of the hemagglutination inhibition (HAI) assay method.
Time Frame: Day 0 and Day 28 post-vaccination
Population: Seroconversion to the vaccine antigens was assessed in the full analysis set population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fluzone® High-Dose Vaccine Group | Fluzone® Vaccine Group
Number analyzed (Participants) | 145 | 151
Percentage of Participants
  A/H1N1: California | 78 | 78
  A/H3N2: Victoria | 89 | 76
  B: Brisbane | 64 | 41

4. Primary Outcome: Percentage of Participants With Seroprotection Before and After Vaccination With Either Fluzone® High-Dose or Fluzone® Vaccine
Description: Seroprotection was defined as a titer ≥ 40 (1/dilution [1/dil]). Serum antibody titers were assessed by means of the hemagglutination inhibition (HAI) assay method.
Time Frame: Day 0 and Day 28 post vaccination
Population: Seroprotection was assessed in the full analysis set population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fluzone® High-Dose Vaccine Group | Fluzone® Vaccine Group
Number analyzed (Participants) | 147 | 152
Percentage of Participants
  A/H1N1: California - Pre-vaccination (N=147, 152) | 50 | 41
  A/H3N2: Victoria - Pre-vaccination (N=147, 152) | 50 | 51
  B: Brisbane - Pre-vaccination (N=147, 152) | 46 | 47
  A/H1N1: California - Post-vaccination (N=145, 151) | 100 | 98
  A/H3N2: Victoria - Post-vaccination (N=145, 151) | 99 | 98
  B: Brisbane - Post-vaccination (N=145, 151) | 97 | 87

5. Secondary Outcome: Number of Participants Reporting Solicited Injection Site or Systemic Reactions After Vaccination With Either Fluzone® High-Dose or Fluzone® Vaccine
Description: Solicited Injection Site Reactions: Pain, Erythema, Swelling, Ecchymosis, and Induration. Solicited Systemic Reactions: Fever, Headache, Malaise, Myalgia, and Shivering
Time Frame: Day 0 through Day 7 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated subjects with available reaction data, safety analysis set population.
Measure: Number; unit: Participants
Arm/Group | Fluzone® High-Dose Vaccine Group | Fluzone® Vaccine Group
Number analyzed (Participants) | 147 | 152
Participants
  Any Injection Site Pain | 112 | 85
  Grad 3 Injection site Pain-Prevents daily activity | 1 | 0
  Any Injection Site Erythema | 11 | 2
  Grade 3 Injection Site Erythema (>100 mm) | 0 | 0
  Any Injection Site Swelling | 9 | 2
  Grade 3 Injection Site Swelling (>100 mm) | 0 | 0
  Any Injection Site Ecchymosis | 1 | 1
  Grade 3 Injection Site Ecchymosis (>100 mm) | 0 | 0
  Any Injection Site Induration | 13 | 3
  Grade 3 Injection Site Induration (>100 mm) | 0 | 0
  Any Fever | 1 | 0
  Grade 3 Fever (≥ 39.0 ºC or ≥ 102.1 ºF) | 0 | 0
  Any Headache | 46 | 40
  Grade 3 Headache (Prevents daily activity) | 5 | 3
  Any Malaise | 44 | 38
  Grade 3 Malaise (Prevents daily activity) | 10 | 5
  Any Myalgia | 70 | 46
  Grade 3 Myalgia (Prevents daily activity) | 10 | 4
  Any Shivering | 29 | 21
  Grade 3 Shivering (Prevents daily activity) | 7 | 3

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination through 28 days post-vaccination.
Arm/Group | Fluzone® High-Dose Vaccine Group | Fluzone® Vaccine Group
Serious Adverse Events (participants affected / at risk) | 0/148 | 0/152
Other Adverse Events (participants affected / at risk) | 130/148 | 110/152
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Fluzone® High-Dose Vaccine Group (N=148) | Fluzone® Vaccine Group (N=152)
Solicited Injection Site Pain (General disorders) | 112 (112) | 85 (85)
Solicited Injection Site Erythema (General disorders) | 11/147 (11) | 2 (2)
Solicited Injection Site Swelling (General disorders) | 9/147 (9) | 2 (2)
Solicited Injection Site Induration (General disorders) | 13/147 (13) | 3 (3)
Solicited Malaise (General disorders) | 44/147 (44) | 38 (38)
Solicited Shivering (General disorders) | 29/147 (29) | 21 (21)
Solicited Myalgia (Musculoskeletal and connective tissue disorders) | 70/147 (70) | 46 (46)
Solicited Headache (Nervous system disorders) | 46/147 (46) | 40 (40)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.